CLINICAL TRIAL: NCT04706832
Title: Thoracic Splanchnic Magnetic Neuromodulation Therapy (ThorS-MagNT) for Grade 3 Diabetic Gastroparesis: Pilot Study
Acronym: ThorS-MagNT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThorS-MagNT; U24DK115255-04 (NIH); U24DK076169-13 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Gastroparesis

STUDY DESIGN:
Intervention Model Description: Intervention type: FDA regulated device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ThorS-MagNT Treatment (Other): Low-frequency, low-intensity repetitive magnetic stimulation bilaterally at T7-8 intravertebral space twice a day for 5 days with a total 1200 magnetic stimulations per treatment session at 1 Hz.
  Interventions: Device: Thoracic Splanchnic Magnetic Neuromodulation Therapy

INTERVENTIONS:
Device: Thoracic Splanchnic Magnetic Neuromodulation Therapy — ThorS-MagNT is performed by low-frequency, low-intensity repetitive magnetic stimulation bilaterally around T7-8 intervertebral space twice a day for 5 days with a total 1200 magnetic stimulations per treatment session at 1 Hz.
  Other Names: ThorS-MagNT

SUMMARY:
Diabetic gastroparesis (DG) is an under recognized and significant complication of diabetes with lack of effective treatments. Recently, a 4-fold increase in hospitalizations has been seen in DG patients with refractory symptoms, defined as Grade 3 gastroparesis. A critical barrier to progress has been both a lack of pathophysiological understanding of DG and absence of effective treatments. Diabetic autonomic neuropathy is felt to be a key dysfunction in DG that causes gastric atony and segmental hypomotility of the small intestine. Autonomic testing of DG patients reveals significant sympathetic hypofunction, a feature distinguishing DG from diabetics with normal gastric emptying. Therefore, stimulation of the thoracic dorsal roots of the greater splanchnic nerve (sympathetic stimulation) could enhance gastric motility, as observed in animal models, and improve DG.

Investigators have developed a novel, safe, noninvasive peripheral nerve treatment using repetitive magnetic stimulation, and have demonstrated improvement in fecal incontinence with neuropathy. The goal of this study is to build on our expertise to conduct a pilot, feasibility study by examining the effect of Thoracic Splanchnic Magnetic Neuromodulation Therapy (ThorS-MagNT) in patients with Grade 3 DG. The aims are to evaluate the safety, effectiveness and feasibility of ThorS-MagNT in patients with Grade 3 DG and to evaluate predictive factors of treatment. The central hypothesis is that ThorS-MagNT will improve sympathetic hypofunction, gastric motility, and spino-gut interactions, and thereby, improve symptoms of DG.

ThorS-MagNT will be performed in 12 patients hospitalized with severe DG by using low-frequency, low-intensity repetitive magnetic stimulation, bilaterally, around T7 intravertebral space, twice a day for 5 days, with a total 1200 magnetic stimulations per treatment session at 1 Hz. The primary outcome is responder rate, defined as ≥20% reduction in the Gastroparesis Cardinal Symptom Index-daily diary (ANMS GCSI-DD) score. Secondary outcomes include subscores of the ANMS GSCI-DD, effects on gastric emptying time, Patient Global Impression of Improvement (PGI-I), safety, and tolerability. The impact of this work is to develop a novel, safe, and non-invasive treatment for severe DG that could result in a paradigm shift in management of DG.

DETAILED DESCRIPTION:
The global burden of diabetes, both type 1 (TIDM) and type 2 (T2DM), is increasing. Gastroparesis is an under-recognized and significant complication of diabetes, whose lack of effective treatment has severely handicapped diabetic management. Diabetic gastroparesis (DG) can range up to half of T1DM patients in tertiary care. Recently, a 4-fold increase in hospitalizations has been seen in DG patients with refractory symptoms despite medical therapy and inability to maintain oral nutrition - Grade 3 gastroparesis or gastric failure. A critical barrier to progress has been both a lack of pathophysiological understanding of DG and absence of effective treatments. A key dysfunction in DG is felt to be diabetic autonomic neuropathy (DAN) that causes gastric atony and segmental hypomotility of the small intestine, in addition to disruption of urinary bladder function, sudomotor, pilomotor, and vasomotor activities. Autonomic testing of DG patients in the NIDDK Gastroparesis Clinical Research Consortium (GpCRC) showed sympathetic hypofunction was the only significant abnormality that distinguished DG from diabetics with normal gastric emptying. The greater splanchnic nerve carries a mix of sympathetic and parasympathetic nerve fibers in the abdomen6. Stimulation of the thoracic dorsal roots or the greater splanchnic nerve in the thorax, pure sympathetic stimulation, may enhance gastric contractility especially in states of gastric atony or hypocontractility, as demonstrated in multiple animal studies.

Investigators have developed a novel, safe, noninvasive, and effective peripheral nerve treatment, translumbosacral neuromodulation therapy (TNT), using repetitive magnetic stimulation, for fecal incontinence (FI). In FI patients, investigators have demonstrated that TNT can correct neuropathy and improve bowel function. The goal of this study is to build on investigators' expertise to conduct a pilot, feasibility study by examining the effect of Thoracic Splanchnic Magnetic Neuromodulation Therapy (ThorS-MagNT) in patients with Grade 3 DG. Central hypothesis is that ThorS-MagNT will improve sympathetic hypofunction, gastric hypomotility/atony, and spino-gut interactions and thereby improve symptoms of DG. The impact of this work is to develop a safe, non-invasive neuromodulation therapy for severe DG.

Specific Aim #1 - Evaluation of the Safety and Effectiveness of Thoracic Splanchnic Magnetic Neuromodulation Therapy (ThorS-MagNT) in patients with Grade 3 Diabetic Gastroparesis. To test the hypothesis that ThorS-MagNT will reduce symptoms of gastroparesis, improve gastric emptying, and is well-tolerated. ThorS-MagNT is performed by low-frequency, low-intensity repetitive magnetic stimulation bilaterally around T7-8 intravertebral space twice a day for 5 days with a total 1200 magnetic stimulations per treatment session at 1 Hz. The primary outcome is responder rate, defined as ≥20% reduction in the Gastroparesis Cardinal Symptom Index-daily diary (ANMS GCSI-DD) score. Secondary outcomes include subscores of the ANMS GSCI-DD, effects on gastric emptying time, Patient Global Impression of Improvement (PGI-I), safety, and tolerability.

Specific Aim #2 - Determination of predictive factors for response to ThorS-MagNT for Diabetic Gastroparesis. To test the hypothesis that subjects with more severe disease as assessed by the Patient Global Impression of Severity (PGI-S), poorly controlled diabetes, increased Brain-derived neurotrophic factor (BDNF), and significant neuroinflammation will predict better response to ThorS-MagNT.

Successful completion of this proposal will establish thoracic splanchnic neuromodulation as a promising, safe, and non-invasive therapy for diabetic gastroparesis, a condition sorely lacking in effective treatments, with potential to induce neuroplastic changes along the spino-gastrointestinal pathway and result in a paradigm and conceptual shift in current management of DG.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed diabetic gastroparesis patients admitted with persistent symptoms after correction of metabolic disturbance;
2. Men or women age less than 85;
3. No known mucosal disease

Exclusion Criteria:

1. Postsurgical gastroparesis;
2. Gastrointestinal obstruction or presence of gastric bezoar;
3. Prior gastric surgery (fundoplication, gastric resection or pyloroplasty);
4. Active inflammatory bowel disease;
5. Eosinophilic gastroenteritis;
6. Connective tissue disease;
7. Chronic liver disease;
8. Use of opioids, tricyclic antidepressants;
9. Active depression;
10. Severe cardiac disease and arrhythmias;
11. Metal implants, including gastric electrical stimulators (GES) deep brain stimulators (DBS), sacral nerve stimulators (SNS), or pacemakers;
12. Pregnant women or nursing mothers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Responder rate | 1 week
  The responder rate is defined as an improvement in the Gastroparesis Cardinal Symptom Index-daily diary (ANMS GCSI-DD) score (e.g., >20% decrease in total symptom score from baseline) in at least 50% of the days of treatment.

SECONDARY OUTCOMES:
Sub-scores of the ANMS GSCI-DD | 1 week
  The change in 1. severity of nausea, 2. severity of early satiety, 3. severity of postprandial fullness, 4. severity of upper abdominal pain, 5. number of vomiting episodes, and 6. severity of gastroparesis during 5 days of ThorS-MagNT treatment.
Gastric emptying time | 3 weeks
  The change in gastric emptying time after 5 days of ThorS-MagNT treatment and 14 days after treatment.
Patient Global Impression of Improvement (PGI-I) | 3 weeks
  The change in Patient Global Impression of Improvement (PGI-I) score after 5 days of ThorS-MagNT treatment and 14 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Sharma, MD, MS, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karunaratne T, Yan Y, Eubanks A, Inman B, Rao S, Sharma A. Thoracic Spinal Nerve Neuromodulation Therapy for Diabetic Gastroparesis: A Proof-of-Concept Study. Clin Gastroenterol Hepatol. 2023 Oct;21(11):2958-2959.e3. doi: 10.1016/j.cgh.2022.09.012. Epub 2022 Sep 22. No abstract available. PMID 36152902